CLINICAL TRIAL: NCT00167297
Title: A Pilot Trial of Atomoxetine to Enhance Motivational Interviewing Therapy for the Treatment of Cannabis Dependence
Brief Title: Atomoxetine for the Treatment of Cannabis Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Kyle Kampman, M.D., University of Pennsylvania, Treatment Reseach Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 801701; P60DA005186-17 (NIH); T32MH019126-14 (NIH); T32MH019126-15 (NIH); T32MH019126-16 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2010-06

CONDITIONS: Cannabis Dependence
Keywords: atomoxetine; cannabis dependence; treatment
MeSH Terms: conditions — Marijuana Abuse | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental): Atomoxetine (Strattera) 25mg peroral (PO) each day for seven days, then up to 40mb bid 40mg PO each day for three days, then 80mg PO bid.
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
The purpose of this small open-label trial is to evaluate the feasibility of recruiting cannabis dependent patients for treatment with Atomoxetine and MIT. The clinical data to date on Atomoxetine has been limited to children and adults with attention deficit disorder without co-morbid substance dependence. However, one study estimated that adults with attention deficit disorder have rates of drug abuse three to four times higher than controls (Mannuzza S 1998). The study also reported that cannabis and cocaine are most frequently abused in this population.

DETAILED DESCRIPTION:
This is a Phase 2 open-label study. We will recruit 10 cannabis dependent subjects and treat them with the combination of Atomoxetine and MIT to reduce their consumption of cannabis. Subjects will be 10 men and women with current DSM-IV diagnosis of cannabis dependence. All patients will receive Atomoxetine and four sessions of MIT. The study length for each patient will be one week for baseline screening and starting medication. This is followed by 8 weeks of medication and an end of study visit one week after completing medications.

The PI will review all information collected regarding the subject's eligibility for the study. The subject will return approximately four days later, and if the PI finds the subject suitable for the study, the subject will begin taking study medication. This visit is referred to as visit 2. During visit 2, the PI will monitor the subject for concomitant medications and adverse events. The research technician will collect Vital Signs, Weight, BAL, the TLFB, a Urine Tox Screen and THC/CR ratio. Both visits 1 and 2 will be conducted within the first week of the study. Starting at visit 2, subjects will take one 25mg capsule of Atomoxetine orally for seven days. Beginning at visit 3, subjects will increase the dose to 40mg per day for 3 days, followed by 80mg (two 40mg capsules concurrently) for the other four days of the second week. Beginning with week 3, subjects will take two 40mg capsules (80mg total) every day of the week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-65 years old
* Meets DSM-IV criteria for Cannabis Dependence
* Live within a commutable distance of the Treatment Research Center
* Understands and signs the informed consent

Exclusion Criteria:

* Current DSM-IV diagnosis of any psychoactive substance dependence other than marijuana, or nicotine dependence
* History of a learning disability
* History of a diagnosis of ADHD made by a psychiatrist.
* Concomitant treatment with psychotropic medications, especially Monoamine Oxidase Inhibitors
* Mandated to treatment based upon a legal decision or as a condition of employment
* Current severe psychiatric symptoms, e.g. psychosis, dementia, acute suicidal or homicidal ideation, mania or depression requiring antidepressant therapy, or which could make it unsafe for the patient to participate in the opinion of the primary investigators.
* Use of any investigational medication within the past 30 days
* Current treatment with pressor agents or albuterol.
* History of narrow angle glaucoma.
* History of significant, unstable heart disease, including myocardial infarction, unstable angina, cardiac failure, second or third degree heart block, or uncontrolled hypertension
* Known hypersensitivity to atomoxetine
* Subjects with known AIDS or other serious illnesses, which may require hospitalization during the study
* Female subjects who are pregnant or lactating, or female subjects of child bearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include:

Barrier (diaphragm or condom) with spermicide Intrauterine device Levonorgestrel implant Medroxyprogesterone acetate contraceptive injection Oral contraceptives

-Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the principal investigators. On EKG, 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed. Liver function tests (LFT's) <5 times ULN without symptoms of liver disease are acceptable after thorough medical review.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Marijuana use in patients treated with atomoxetine and Motivational Interviewing Therapy measured using weekly urine drug screens. | 8 weeks

SECONDARY OUTCOMES:
Tolerability of atomoxetine: Tolerability will be assessed by examining the rates of certain adverse events during the treatment phase. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlos F. Tirado, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Rersearch Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Tirado CF, Goldman M, Lynch K, Kampman KM, Obrien CP. Atomoxetine for treatment of marijuana dependence: a report on the efficacy and high incidence of gastrointestinal adverse events in a pilot study. Drug Alcohol Depend. 2008 Apr 1;94(1-3):254-7. doi: 10.1016/j.drugalcdep.2007.10.020. Epub 2008 Jan 7. PMID 18182254